CLINICAL TRIAL: NCT04149561
Title: Evaluation of Communication Functions in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: BVUFTRCP1
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; communication
MeSH Terms: conditions — Cerebral Palsy; Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cerebral Palsy: 100 patients over 2 years of age with a diagnosis of cerebral palsy will be included in the study. Demographic information form prepared for the study in terms of demographic information such as age, gender, clinical type of cerebral palsy, drugs used, comorbid diseases will be completed. Communication Function Classification System and Functional Communication Classification System will be used to evaluate patients' communication skills. In addition, patients; The Gross Motor Function Classification System for cerebral palsy and based on child-initiated movements with emphasis on sitting, displacement and mobility, and to hold objects during the daily activities of children with cerebral palsy. The Manual Ability Classification System, which classifies how they use their hands, will also be completed.
  Interventions: Other: communication skill measurement with self report questionnaire

INTERVENTIONS:
Other: communication skill measurement with self report questionnaire — Demographic information form, Communication Function Classification System, Functional Communication Classification System, The Gross Motor Function Classification System and Manual Ability Classification System will be filled in for the patients.

SUMMARY:
In this study, investigators aimed to evaluate the communication functions of children between 2-18 with cerebral palsy. Investigators planned to investigate the relationship between communication skills and clinical characteristics and socio-demographic status of the family.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a non-progressive, movement-limiting loss of permanent motor function, posture and movement disturbance in the developing brain due to lesion or injury that occurs during the intrauterine period or in the first months of life. Secondary medical problems such as epilepsy, mental retardation, behavior disorder, swallowing problems and musculoskeletal disorders may be seen in these patients. Neuroanatomical problems in the muscles associated with the mouth and speech, and the presence of central pathologies, are important problems in patients with cerebral palsy. Monitoring the communication level of these patients is very important for determining treatment protocols and monitoring their effectiveness. Difficulties in communication significantly affect the rate and level of recovery in patients with cerebral palsy. There are many different scales to analyze communication level and problems in children with cerebral palsy. The most commonly used ones are the Communication Function Classification System (CFCS) and the Functional Communication Classification System (FCCS). By examining the communication level in 5 categories in both scales, it helps to monitor the communicative development of the child and also provides a common language among clinicians. They are defined by the World Health Organization (WHO) and focus on the levels of activity and participation defined in the international classification of function, disability and health.

The aim of this study was to evaluate the communication level in children over 2 years of age with cerebral palsy. In addition, the relationship between communication skills and general functional levels and demographic characteristics will be investigated. In this way, both the general communication level of this patient group and the possible factors affecting this skill will be analyzed. Thus, these relationships and measurements can be utilized in determining treatment and rehabilitation protocols.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose parents agreed to participate in the study.
* Patients with confirmed cerebral palsy.
* Patients aged 2-18 years.

Exclusion Criteria:

* Patients without definite cerebral palsy.
* Patients whose family refused to participate in the study.
* Patients with another neurological disorder that may affect their physical and neurological capacity.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 100 patients aged 2-18 years with cerebral palsy.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-03-14 (Actual)

PRIMARY OUTCOMES:
Functional Communication Classification System(FCCS) | 6 month
  The Functional Communication Classification System was designed to classify how children with cerebral palsy between the ages of four and five communicate on a daily basis. The tool focuses on how children typically communicate with familiar and unfamiliar communication partners. There are five classifications a child can be categorized in: (1) effective communicator in most situations (2) effective communicator in most situations, but does need some help (3) an effective communicator in most situations and can communicate small ranges of messages and topics to most familiar people (4) assistance is required in most situations, especially with unfamiliar people and environments. Communicates daily needs and wants to familiar people (5) communicates using undirected movement, vocalisation and/or behaviour, for interpretation by familiar people.
Communication Function Classification System (CFCS) | 6 month
  The CFCS is a tool used to classify the everyday communication of an individual with cerebral palsy into one of five levels according to effectiveness of communication. It consists of five levels which describe everyday communication ability.
  Classification on the CFCS is made by a person who is familiar with the individual's communication in everyday situations.
  Classification is based on the effectiveness of communication between a sender and receiver of information.
  CFCS considers the familiarity of a person's communication partners.
  All ways of communicating are considered including speech, gesture, facial expression and augmentative and alternative communication.
  A person classified at Level I is a more able communicator than a person classified at Level V.
Gross Motor Function Classification System (GMFCS) | 6 month
  The Gross Motor Function Classification System (GMFCS) for cerebral palsy is based on self-initiated movement, with emphasis on sitting, transfers, and mobility. When defining a five-level classification system, our primary criterion has been that the distinctions between levels must be meaningful in daily life. Distinctions are based on functional limitations, the need for hand-held mobility devices (such as walkers, crutches, or canes) or wheeled mobility, and to a much lesser extent, quality of movement. The distinctions between Levels I and II are not as pronounced as the distinctions between the other levels, particularly for infants less than 2 years of age.
Manual Ability Classification System (MACS) | 6 month
  The Manual Ability Classification System (MACS) describes how children with cerebral palsy use their hands to handle objects in daily activities. MACS describes five levels. The levels are based on the children's self-initiated ability to handle objects and their need for assistance or adaptation to perform manual activities in everyday life.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif university, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No